CLINICAL TRIAL: NCT05868798
Title: Effects of 36 Hours of Sleep Deprivation on Military-related Tasks: Can Ammonium Inhalants Maintain Performance?
Brief Title: Can Ammonium Inhalants Maintain Performance in Sleep Deprived Soldiers?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jan Malecek (Other)
Responsible Party: Sponsor-Investigator, Jan Malecek, Principal Investigator, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SleepStudy01
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Sleep Deprivation; Military Activity; Sleep; Cognitive Change; Military Combat Stress Reaction
Keywords: cognition; military; sleep deprivation; performance; ammonia
MeSH Terms: conditions — Sleep Deprivation | interventions — Ammonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants performed each individual test without ammonia inhalants.
- Ammonia inhalants (Experimental): Participants performed each individual test with ammonia inhalants.
  Interventions: Drug: Ammonia Inhalant

INTERVENTIONS:
Drug: Ammonia Inhalant — For all AI trials, a capsule containing 0.3 mL of AI (composed of 15% of ammonia and 35% of alcohol) was used according to the manufacturer's instructions (Dynarex Corporation, Orangeburg, NY). When the ammonia fumes were released, researcher immediately held the capsule under the participant's nose to inhale until a voluntary withdrawal reflex was observed.
  Other Names: smelling salt
  Arms: Ammonia inhalants

SUMMARY:
This study aims to examine the effectiveness of ammonia inhalants in countering the effects of total sleep deprivation on cognitive and physical performance tests relevant to military personnel.

DETAILED DESCRIPTION:
Data from this study are part of a broader research project aimed at investigating the effects of different light conditions on cognitive and physiological performance during periods of total sleep deprivation. We used a crossover randomized controlled trial design with within-subject repeated-measures to assess the effects of ~36 hours of total sleep deprivation and acute ammonia inhalation on occupationally relevant military tasks in military personnel.

Participants reported to the Sleep and Chronobiology laboratory (National Institute of Mental Health) on Thursday evening after a standardized dinner at ~1800 h. They then completed a series of questionnaires addressing psychological and physiological health, which were followed by a general familiarization of the layout of the facility (i.e., location of the bathrooms, testing stations, etc.). During this familiarization, the participants were also familiarized with the specific testing procedures and practiced each of the required tasks.

The actual testing protocol began with a night of uninterrupted sleep from ~2200 h to ~0630 h. Participants then underwent 5 identical testing sessions from every ~0730-0930 h in the morning and ~1900-2100 h in the evening. The first test occurred in the morning after the full night of baseline sleep (0 h) and again after 12 hours (-12 h), 24 hours (-24 h), and 36 hours of total sleep deprivation (-36 h) followed by additional testing session after 8 hours (from 2230-0630 h) of recovery sleep (+8 h). During total sleep deprivation, participants were not allowed to sleep and were kept awake in a common room by passive means, such as playing board games, watching television and reading books while under constant supervision of the research team. Furthermore, the participants were subjected to a constant ambient room light for the entire duration of total sleep deprivation period.

Participants were administered a standardized sleepiness scale and underwent simple reaction time testing, handgun shooting accuracy protocol, a rifle disassembly and reassembly protocol, and countermovement jump testing at each testing session. Participants performed each individual test twice at each testing period, either with AI (AI) or without AI (CON), in randomized order and separated by 2 minutes of rest (in order to minimize any potential carryover effects of the AI)

For all AI trials, a capsule containing 0.3 mL of AI (composed of 15% of ammonia and 35% of alcohol) (31) was used according to the manufacturer's instructions (Dynarex Corporation, Orangeburg, NY). When the ammonia fumes were released, researcher immediately held the capsule under the participant's nose to inhale until a voluntary withdrawal reflex was observed.

During the entire study protocol, participants received personalized daily food rations consisting of standard 'ready to eat' meals commonly used in the Czech military. One week before the experiment, participants' body composition was measured (using air displacement plethysmography; Bod Pod Body Composition System; Life Measurement Instruments, Concord, CA), and the total daily energy expenditure was derived from the estimated resting metabolic rate and application of an "active" physical activity factor of 1.6 to the individual caloric requirements. In addition, each participant was allowed ad libitum water consumption. Breakfast was consumed at ~0930 h, lunch at ~1230 h, and dinner at ~1730 h, each day. Additionally, all forms of stimulants were prohibited 72 hours before and during the testing protocol.

ELIGIBILITY:
Inclusion Criteria:

* passed an annual physical fitness test
* passed medical checkup within the last year
* have at least two years of active-duty service experience
* report a high level of comfort handling firearms
* non-smokers
* currently not working shift-work
* not taking medications known to interfere with sleep, cognitive or physical performance.

Exclusion Criteria:

* smoker
* did not pass an annual physical fitness test
* did not pass medical checkup within the last year
* work in Shift-work

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The cadets were selected (Q1, 2021) primarily due to their homogenous (this brach of study now study only men) and synchronized daily cycle based on mandatory morning lineups and the University program.
Enrollment: 18 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Epworth sleepiness scale from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  We used Epworth Sleepiness Scale (ESS) translated into Czech. It is a self-administered eight-item questionnaire and takes two to three minutes to complete. The questionnaire presents daily lifestyle activities (i.e. reading, watching TV etc.) and participants rate their current self-perceived likelihood of dozing off in each situation, from: "would never doze" (0) to "high chance of dozing". The ESS provides a cumulative score between 0 and 24, with higher numbers indicating greater sleepiness.
Change in simple reaction time from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  A simple reaction time test was used to assess the speed of responses to visual stimuli. The evaluation of reaction time was performed using the PEBL Version 2.0 software. The test consists of instantaneous responses to a visual stimulus by pressing a spacebar key on a laptop's keyboard as quickly as possible when a visual stimulus appears. In the test, 50 trials of stimuli were presented with an interstimulus interval that randomly varied between 250 ms and 2500 ms. Each participant completed four tests (each time two, either with AI or CON, in randomized order) with 2 minutes of inter-test rest. The simple reaction time data obtained were inspected according to pre-determined criteria, which excluded trial executions that were deemed incorrect due to a reaction time shorter than 150 ms or longer than 3000 ms. The mean reaction time (measured in milliseconds) and the number of incorrect trial executions were used as the variables in the subsequent statistical analysis.
Change in handgun shooting accuracy from baseline | Performed in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  A laser-based simulator system with an infrared laser handgun was used to assess handgun shooting accuracy. All trials were performed in the standardized isosceles high-ready stance position. For this study, a real-weight mock-up of the Czech military standard issue Glock 17/22 handgun was used (all participants were familiar with the handgun from their active service). Participants wore over-ear headphones during all testing procedures to hear the software command to start shooting and the simulated shooting blasts when pulling the trigger. A 20 cm circular target was placed on a blank wall 4 meters in front of the participants to simulate a standard-issue 50 cm target 10 meters away for the laser-based handgun shooting protocols. For the testing, participants fired 10 shots, aiming to hit the middle of the circular target (a bullseye hit was worth 10 points, and 1 point was deducted for every 1 cm region away from the bullseye, resulting in a maximum score of 100 points).
Change in rifle disassembling and reassembling from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  The protocol for disassembling and reassembling a military-standard issue assault rifle was selected to assess changes in manual dexterity as it is representative tasks that soldiers may encounter in field operations. During the protocol, participants were tasked to disassemble and reassemble a rifle consisting of 8 parts as fast as possible. Prior to the task's onset, standing participants were instructed to place their hands behind their backs and wait for the researcher's "start" command, after which they attempted to disassemble the rifle as quickly as possible. After a two-minute break, during which participants organized the rifle parts on a table, they then proceeded to reassemble the rifle under the same instruction, and the time was recorded. During the reassembling, the final step was conducting a successful "rifle function check". The time for completion of the task was measured using a handheld stopwatch and recorded on a digital camera for possible corrections.
Change in countermovement jump height from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  We used unloaded countermovement jump (CMJ), one of the most common and straightforward strategies to monitor short-term neuromuscular performance in tactical populations. Each CMJ session included 2 sets (AI and CON in a randomized order) of 3 maximal effort CMJs with 2 min of inter-set standing rest. The researcher verbally instructed and encouraged the participants to jump as high as possible on each jump. All CMJs were performed with wooden dowel (~ 0.5 kg) as a mock barbell placed across the participant's upper back mimicking a regular back squat. A linear position transducer (GymAware Power Tool; Kinetic Performance Technologies, Canberra, Australia) was attached to both sides of a dowel to measure the performance. The depth of the CMJ depth was self-selected. Participants wore the same sports t-shirts, shorts and shoes during each test period. The mean of the 3 jump heights (cm) was calculated for each condition at each test session.
Change in heart rate from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  All participants wore a chest strap heart rate monitor (Polar Electro Inc., Model H10, Lake Success, NY, USA) during the shooting protocol. Baseline heart rate data were derived as a mean of heart rate from 2 minutes immediately preceding the start of the shooting trial. Heart rate (bpm) was then continuously monitored during all sessions of shooting protocol. After baseline testing, heart rate data were averaged in 15 seconds bins (0-15, 15-30, 30-45, 45-60) for one minute immediately following the AI and CON trials. The mean of these bins from each trial was used in subsequent analysis.
Change in rating of perceived exertion from baseline | We were following changes in 5 identical testing sessions during 36 hours of total sleep deprivation (after 0-baseline, 12, 24, and 36 hours), and after 8 hours of recovery sleep.
  The rating of perceived exertion (RPE) was recorded during the CMJ testing using a CR-10 scale to evaluate RPE scores after each set of CMJ. RPE is a frequently used marker of exercise intensity typically used for monitoring during exercise tests to complement other intensity measures.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malecek, Principal Investigator — Faculty of Physical Education and Sport, Charles University, Prague, Czech Republic
Locations (1):
- Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After manuscript publication.
Access Criteria: Individuals' data will only be provided to them on request and on proof of their identity.